CLINICAL TRIAL: NCT04534673
Title: Pegylated Interferon Lambda for Treatment of COVID-19 Infection- A Randomized Open Label Pilot Trial
Brief Title: Pegylated Interferon Lambda for Treatment of COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ohad Etzion, Director, Department of Gastroenterology & Liver Diseases, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0129-20-SOR; SCRC200006 (Other: Soroka Clinical Research Center)
Record Dates: First submitted 2020-04-20; First posted 2020-09-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Pegylated interferon lambda
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A randomized, open label, 2 arm, pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pegylated interferon lambda + Standard of care treatment
  Interventions: Drug: Lambda 180 mcg S.C
- Control group (No Intervention): Standard of care treatment

INTERVENTIONS:
Drug: Lambda 180 mcg S.C — Prefilled injection syringe of 180 microgram Pegylated interferon lambda, administered on day 0 and if needed on day 7
  Other Names: Lambda
  Arms: Intervention group

SUMMARY:
A randomized, open-label, 2 arm, pilot trial of Lambda 180 mcg administered subcutaneously once weekly, for up to two weeks (2 injections at most), in addition to standard supportive care, compared to standard supportive care alone, in a population of COVID-19 infected patients.

patients will be randomized according to 1:1 ratio to one of the 2 trial arms: Lambda 180 mcg S.C + standard care (intervention arm) or standard care only (control arm).

DETAILED DESCRIPTION:
Recently, a novel coronavirus (SARS-CoV-2) has been identified as the causative pathogen of a rapidly spreading infection associated with pneumonia and severe acute respiratory syndrome (COVID-19), for which there is currently no approved therapy. Interferon Lambda (IFN Lambda) is a type III interferon with broad anti-viral activity and receptor distribution limited to the respiratory and gastrointestinal epithelium. Studies in animal models suggest that IFN Lambda may ameliorate infection with respiratory viruses such as influenza coronaviruses. The WHO has recently included pegylated interferon lambda in its landscape analysis of potential therapeutics for COVID-19.

In this randomized, open-label, 2 arms, pilot trial, up to 40 patients diagnosed with COVID-19 and mild to moderate respiratory infection, will be randomized to one of 2 treatment arms in 1:1 ratio: 1. Lambda 180 mcg administered S.C once weekly, for up to two weeks (2 injections at most) + standard care, Or 2. Standard care alone.

Efficacy of Lambda will be assessed by PCR analysis for COVID-19 (Fluxergy, Irvine CA), from respiratory secretions obtained by nasopharyngeal and oropharyngeal swabs, collected consecutively at day 1, 3, 5, 7, 10, 14 and 21 following initial diagnosis or until patients are discharged following achievement of two consecutive PCR negative tests for COVID-19. Safety and tolerability of Lambda will be assessed by adverse event (AE) monitoring, vital signs assessment and clinical laboratory tests (CBC, and extended chemistry panel).

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients over the age of 18.
2. Confirmed COVID-19 infection by PCR analysis
3. Hospitalized at Soroka University Medical Center.
4. Display mild to moderate symptoms of respiratory infection (Temperature <39.0 oC, respiratory rate < 25, O2 % Sat > 95% in room air or with supplemental oxygen through nasal cannula, P/F ratio > 150).
5. Willing and able to convey informed consent.
6. Willing and able to comply with all study procedures
7. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal.

For females: 2 of the following contraceptive methods, with at least 1 being a barrier method:

* Hormonal contraceptives for ≥ 27 days before dosing
* Intrauterine device (IUD) in place ≥ 27 days before dosing
* Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening
* Surgical sterilization of the partner (vasectomy ≥ 1 month before screening) Female patients must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of investigational product.

For males:

* Surgical sterilization (vasectomy ≥ 1 month before screening) Or
* Both of the following contraceptive methods from screening:

  * Consistently and correctly use a condom
  * Partner must use a hormonal contraceptive or a nonhormonal barrier method (IUD or diaphragm with spermicide or cervical cap with spermicide).

Exclusion Criteria:

1. Treatment with interferons (IFNs) immunomodulators and/or immunosuppressive or B-cell depleting medications within 12 months before screening.
2. Previous use of Interferon Lambda. Patients who previously participated in a clinical trial of Interferon Lambda but are confirmed to have received placebo or another non-Lambda IFNs are allowed.
3. History or evidence of any intolerance or hypersensitivity to IFNs.
4. Patients with respiratory infection requiring invasive or non-invasive ventilatory support (bipap or intubation and mechanical ventilation).
5. Participation in a clinical trial with use of any investigational drug within 30 days before screening.
6. History of any of the following diseases or conditions:

   * Advanced or decompensated liver disease (presence or history of bleeding varices, ascites, encephalopathy or hepato-renal syndrome)
   * Immunologically mediated disease (e.g., rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) that requires more than intermittent nonsteroidal anti-inflammatory medications for management or that requires use of systemic corticosteroids in the 6 months before screening (inhaled asthma medications are allowed).
   * Retinal disorder or clinically relevant ophthalmic disorder.
   * Any malignancy within 5 years before screening. Exceptions are superficial dermatologic malignancies (e.g., squamous cell or basal cell skin cancer treated with curative intent).
   * Cardiomyopathy, significant ischemic cardiac or cerebrovascular disease (including history of angina, myocardial infarction, or interventional procedure for coronary artery disease), or cardiac rhythm disorder.
   * Chronic pulmonary disease (e.g., chronic obstructive pulmonary disease) associated with functional impairment.
   * Pancreatitis.
   * Severe or uncontrolled psychiatric disorder, e.g., depression, manic condition, psychosis, acute and/or chronic cognitive dysfunction, suicidal behavior, and relapse of substance abuse.
   * Active seizure disorder defined by either an untreated seizure disorder or continued seizure activity within the preceding year despite treatment with anti-seizure medication.
   * Bone marrow or solid organ transplantation
   * Other significant medical condition that may require intervention during the trial (such as uncontrolled diabetes or thyroid disease) Patients with any serious condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed. Patients for whom participation in the trial would increase their risk.
   * Current eating disorder
   * Current alcohol abuse (excessive alcohol intake, defined as follows: >20 g/day for females [1.5 standard alcohol drinks] or >30 g/day for males [2.0 standard alcohol drinks]. A standard drink contains 14 g of alcohol: 360 mL of beer, 150 mL of wine, or 45 mL of spirits
   * Drug abuse within the previous 6 months before screening, with the exception of cannabinoids and their derivatives
7. Any of the following abnormal laboratory test in the 12 months prior to enrollment

   * Platelet count <90,000 cells/mm3
   * White blood cell (WBC) count <3,000 cells/mm3
   * Absolute neutrophil count (ANC) <1,500 cells/mm3
   * Hemoglobin <11 g/dL for women and <12 g/dL for men
   * Estimated creatinine clearance (CrCl) < 50 mL/min by Cockroft-Gault formulation
   * ALT and/or ALT levels > 10 times the upper limit of normal
   * Bilirubin level ≥ 2.5 mg/dL unless due to Gilbert's syndrome
   * Serum albumin level <3.5 g/dL
   * International normalized ratio (INR) ≥1.5 (except patients maintained on anticoagulant medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Viral shedding in days since initial diagnosis | 21 days
  The duration of viral shedding in days since initial diagnosis, as determined by RT-PCR to COVID-19.
Rate of adverse events and severe adverse events | 21 days from entry
  Rate of treatment-emergent and treatment-related severe adverse events (SAEs)

SECONDARY OUTCOMES:
Time to clinical recovery | 72 Hours
  the time (in hours) from initiation of trial treatment (Lambda or standard care) until normalization of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 72 hours.
Rate of non-invasive or mechanical ventilation | 28 Days
  Requirement for non-invasive (bipap) or mechanical ventilation
Length of hospital stay | 28 Days
  length of hospital stay from admission to discharge
All-cause mortality | At day 28 following admission to the hospital
  All-cause mortality
Undetectable COVID-19 virus levels | At days 7,14 and 21 from admission
  Rate of undetectable COVID-19 virus levels at different days

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Etzion, MD, Principal Investigator — Soroka Univeersity Medical Center
Locations (1):
- Soroka UMC, Beersheba, Israel